CLINICAL TRIAL: NCT05003037
Title: A Open-label, Single Center, Phase II Study of Surufatinib Combined With Toripalimab and Chemotherapy in Patients With Advanced Non-squamous Non-small-cell Lung Cancer
Brief Title: Surufatinib Combined With Toripalimab and Chemotherapy in the Treatment of Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Zhang, MD (Other)
Responsible Party: Sponsor-Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-L102
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wild-type Genotype (Experimental)
  Interventions: Drug: Surufatinib,Toripalimab,Pemetrexed,Carboplatin/Cisplatin
- EGFR mutation (Experimental)
  Interventions: Drug: Surufatinib,Toripalimab,Pemetrexed,Carboplatin/Cisplatin

INTERVENTIONS:
Drug: Surufatinib,Toripalimab,Pemetrexed,Carboplatin/Cisplatin — Surufatinib at the dose determined in phase safety lead-in，250 mg，qd，po，every 3 weeks(q3w) ; Toripalimab at the dose 240mg，iv, d1, given every 3 weeks (q3w); Pemetrexed at the dose 500 mg/m2，iv，d1，given every 3 weeks (q3w); Carboplatin at the dose AUC=5~6，iv，d1，given every 3 weeks (q3w) or Cisplatin at the dose 75 mg/m2，iv ,d1，q3w; Maintenance treatment：After the end of the first-line treatment, patients with CR, PR, and SD can continue to maintenance treatment with Surufatinib RP2D，d1-21，q3w＋Toripalimab 240mg，d1，q3w+Pemetrexed 500mg/m2，d1，q3w was taken until the disease progressed.

SUMMARY:
A phase II study to assess the efficacy and safety of Surufatinib Combined With Toripalimab and Chemotherapy as a first-line treatment in patients with advanced non-squamous non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary provision of informed consent.
2. Males or females aged 18-75.
3. Histological or cytologically confirmed NSCLC, metastatic or non-resectable (stage IIIB-Ⅳ).
4. At least one lesion can be measured by imaging.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
6. Life expectancy ≥ 12 weeks.
7. None previous chemotherapy or targeted therapy(Arm:wild-type genotype).
8. Patients should be confirmed acquired EGFR T790M mutation and received adequate EGFR-TKI treatment(Arm:EGFR mutation).
9. Female of childbearing age must have a negative pregnancy test (serum or urine) within 7 days before enrolment.

Exclusion Criteria:

1. Histological or cytologically confirmed small cell lung cancer (SCLC), including lung cancer mixed with SCLC and NSCLC.
2. Diagnosed with other malignant diseases other than NSCLC within 5 years.
3. Have participated in other interventional clinical research treatments now or within 4 weeks.
4. Have previously received multi-targeted kinase inhibitors therapy.
5. Have active autoimmune diseases requiring systemic treatment within 2 years.
6. Received systemic glucocorticoid therapy or immunosuppressive therapy within 2 weeks.
7. Clinically uncontrollable pleural effusion/abdominal effusion.
8. Vaccinated vaccines or attenuated vaccines within 4 weeks before the group;
9. Pregnant or breastfeeding females.
10. Other serious hazards to the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | up to 24 months

SECONDARY OUTCOMES:
Objective response rate(ORR) | up to 24 months
Disease control rate(DCR) | up to 24 months
Overall Survival(OS) | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China